CLINICAL TRIAL: NCT05138263
Title: Korean Brain Aging Study for Early Diagnosis and Prediction of Alzheimer's disease2
Brief Title: Korean Brain Aging Study for Early Diagnosis and Prediction of Alzheimer's disease2 (KBASE2)
Acronym: KBASE2
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Dong Young Lee, professor, Seoul National University Hospital
Other Study IDs: KBASE02; U01AG072177 (NIH)
Record Dates: First submitted 2021-10-23; First posted 2021-11-30 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment
Keywords: Alzheimer Disease; Early diagnosis; Prediction; Biomarker; Neuroimaging; Network-based analysis; Multiomics; Systems biology
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, Serum, DNA, RNA, hair, and stool
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Young normal controls: * age : 20 ~ 54
  * without dementia, MCI, or other major neurological/psychiatric illness
- Elderly normal controls: * age : 55 ~ 90
  * without dementia, MCI, or other major neurological/psychiatric illness
- MCI (Mild cognitive impairment): * age : 55 ~ 90
  * without major neurological/psychiatric illness
  * concern regarding a change in cognition, lower performance in any cognitive domain that is greater than would be expected for the subject's age and educational background and preservation of independence in functional abilities
- AD (Alzheimer's diseases): * age: 55 ~ 90
  * National Institute of Aging and the Alzheimer's Association (NIA-AA) Probable AD dementia(Alzheimer's diseases)

SUMMARY:
The KBASE2 is the second phase of the KBASE project, which consists of roll-over participants from the first phase of the KBASE as well as newly enrolled participants with varying degrees of cognitive functions (e.g. individuals with normal cognition, mild cognitive impairment, or AD dementia). In addition to the aims of the first phase of the KBASE, the KBASE2 will focus on new data collection and integrative analysis of the rich structural, functional, and molecular neuroimaging data in relation to whole genome sequencing and other -omics. Network analysis of disruption in brain connectivity in relation to clinical status and AD biomarker profiles also will be conducted.

DETAILED DESCRIPTION:
The Korean Brain Aging Study for the Early Diagnosis and Prediction of AD (KBASE) is a comprehensive prospective cohort study launched at Seoul National University (SNU) in 2014 using similar methods to the North American AD Neuroimaging Initiative (ADNI). KBASE includes well-characterized participants with normal cognition (CN), mild cognitive impairment (MCI) and AD dementia. Clinical/cognitive and lifestyle data, multimodal neuroimaging (structural MRI, MR angiography, diffusion tensor imaging, and resting-state fMRI, as well as amyloid, tau and FDG-PET, and bio-specimens were longitudinally collected during the past five years.

The KBASE2, the second phase of the KBASE project, will focus on new data collection and integrative analysis of the rich structural, functional, and molecular neuroimaging data in relation to WGS and other -omics. Network analysis of disruption in brain connectivity in relation to clinical status and AD biomarker profiles in KBASE will be related back to the NIA AD Sequencing Project (ADSP) multi-ethnic dataset (N>20,000) results. Amyloid, tau, neurodegeneration, and cerebrovascular integrity (A/T/N/V) neuroimaging biomarkers will be investigated cross-sectionally and longitudinally. Findings will be contrasted with and validated in independent cohorts, including ADNI and the Indiana Memory and Aging Study (IMAS), which both have similar genetic and deep longitudinal endophenotype data. The overarching premise is that 1) development of precision medicine for ADRD requires systematic multi-modal biomarker collection in diverse cohorts during early at-risk stages of disease to identify diagnostic, prognostic and therapeutic targets, and 2) sophisticated analytic strategies are required to address the complexity of multimodal data, heterogeneity, and diverse participant cohorts. Integrative longitudinal analysis of genetic and -omics networks with structural and functional brain networks in this Asian cohort will yield new targets related to A/T/N/V pathology and other pathways

In KBASE2 projects, the KBASE team at Seoul National University (SNU) and AD research team at Indiana University (ADNI Genetics Core, Indiana ADRC, IU Network Science Institute) will closely collaborate with the ADSP and its multi-institutional working groups, and the Universities of Pennsylvania and Southern California. Whole genome sequences (WGS) will be ADSP-harmonized by the NIA Genomic Center for AD (GCAD) and shared via NIAGADS (both UPenn). The Laboratory of Neuroimaging (LONI; USC) will support imaging and related data sharing.

ELIGIBILITY:
Participants will be classified as either Alzheimer's disease(AD) group, mild cognitive impairment(MCI) group, elderly normal controls or young normal controls. Specific inclusion criteria for each group is described below.

Inclusion Criteria:

[Inclusion criteria: AD]

* Age : 55 - 90
* Clinical Dementia Rating (CDR)=0.5 or 1
* Diagnostic and Statistical Manual-IV(DSM-IV) criteria for dementia
* National Institute of Aging and the Alzheimer's Association (NIA-AA) Probable AD dementia
* Study partner or caregiver to accompany patient to all scheduled visits
* Written informed consent

[Inclusion criteria: MCI (amnestic)]

* Age : 55 - 90
* Clinical Dementia Rating (CDR)=0.5
* Concern regarding a change in cognition (obtained from the subject, from an informant who knows the subject, or from a skilled clinician observing the subject)
* Lower performance in any cognitive domain that is greater than would be expected for the subject's age and educational background
* Preservation of independence in functional abilities
* Study partner or caregiver to accompany subject to all scheduled visits
* Written informed consent

[Inclusion criteria: Elderly normal controls]

* Age : 55 - 90
* Clinical Dementia Rating (CDR)=0
* Those with contactable Informant
* Written informed consent

[Inclusion criteria: Young normal controls]

* Age : 20 - 54
* Clinical Dementia Rating (CDR)=0
* Written informed consent

Exclusion Criteria:

[Exclusion criteria: general]

* Past history or presence of major psychiatric illness (e.g. schizophrenia, bipolar disorder, alcohol/substance abuse or dependence, delirium)
* Significant neurologic or medical condition that can influence the mental state
* Contraindications for MRI scan (e.g. pacemaker, claustrophobia)
* Illiteracy
* Significant visual or hearing difficulty
* Taking investigational drug
* In pregnancy or breast-feeding

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Young and elderly normal controls: community-based population AD and MCI: clinic or community-based population
Sampling Method: Non-Probability Sample
Enrollment: 640 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Amount of brain amyloid deposition | baseline
  Group difference in baseline brain amyloid deposition on florbetaben PET and the relationship between the amount of brain amyloid deposition and clinical, neuropsychological, neuroimaging, genetic, biochemical measurement will be investigated.
Amount of brain tau deposition | baseline
  Group difference in baseline brain amyloid deposition on AV1451 PET and the relationship between the amount of brain tau deposition and clinical, neuropsychological, neuroimaging, genetic, biochemical measurement will be investigated.

SECONDARY OUTCOMES:
Change of brain amyloid deposition | 2 years
  The change of brain amyloid deposition and its relation to the clinical, neuropsychological, neuroimaging, genetic and biochemical variables will be assessed.
Change of brain tau deposition | 2 years
  The change of brain tau deposition and its relation to the clinical, neuropsychological, neuroimaging, genetic and biochemical variables will be assessed.
Change of CERAD total score | 2 years
  The change of CERAD total score and its relation to neuroimaging, genetic and biochemical variables will be assessed.
Change of cortical thickness | 2 years
  The change of Alzheimer-signature region cortical thickness and its relation to neuroimaging, biochemical, genetic biomarkers will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Dong Young Lee, MD, PhD, Principal Investigator — Department of Psychiatry, Seoul National University Hospital
Locations (2):
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - SMG-SNU Boramae Medical Center, Seoul